CLINICAL TRIAL: NCT01671592
Title: Safety and Feasibility Evaluation of the MRI-based Tracking of Alpha-type-1 Dendritic Cell Vaccines in Patients With Colorectal Cancer
Brief Title: Safety of Labeled Dendritic Cell (DC) Vaccines and Feasibility of Tracking by Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pawel Kalinski (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Pawel Kalinski, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-052; R01CA134633 (NIH)
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: Cancer; colorectal; tumor; neoplasms; carcinoma; vaccine
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Carcinoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Day 1 MRI with low dose vaccine (Experimental): DC vaccine at 3 x 10e6 per course which consists of 3 daily intradermal doses per course with the MRI on day 1 of the course.
  Interventions: Biological: DC Vaccine
- Day 3 MRI with low dose vaccine (Experimental): DC vaccine at 3 x 10e6 per course which consists of 3 daily intradermal doses per course with the MRI on day 3 of the course.
  Interventions: Biological: DC Vaccine
- Day 1 MRI with high dose vaccine (Experimental): DC vaccine at 3 x 10e7 per course which consists of 3 daily intradermal doses per course with the MRI on day 1 of the course.
  Interventions: Biological: DC Vaccine
- Day 3 MRI with high dose vaccine (Experimental): DC vaccine at 3 x 10e7 per course which consists of 3 daily intradermal doses per course with the MRI on day 3 of the course.
  Interventions: Biological: DC Vaccine

INTERVENTIONS:
Biological: DC Vaccine — Alpha-type-1-polarized dendritic cells (αDC1) pulsed with apoptotic autologous tumor.

SUMMARY:
This study will evaluate the safety and feasibility MRI tracking of a vaccine produced from a persons cancer cells injected intradermally once a day for 3 consecutive days. One of the daily doses will contain a chemical that can be detected by an MRI. That will be either the 1st or 3rd day of the 3 day course. On that day MRI scans will be performed 6 and 24 hours after the injection on that day. Patients may be able to receive booster doses every 1-2 months

DETAILED DESCRIPTION:
STUDY EVALUATIONS

* Pre-Vaccination

  * Complete physical examination (with ECOG performance status (PS), medical history, weight, height, and BSA); the exact size and location of all tumor lesions will be noted in the flow sheet, documented in the text note, and by photographic and/or radiologic means
  * CEA levels in the blood (as a tumor marker)
  * Women of childbearing potential will have a serum beta-HCG pregnancy test
  * Anti-HIV, HbsAg and Anti-HCV
  * CBC, platelet, differential
  * Comprehensive metabolic panel (CMP) including: glucose, BUN, creatinine, sodium, potassium, Cl, CO2, calcium, total protein, albumin, alkaline phosphatase, AST, ALT, total bilirubin
  * PT/PTT testing
  * Electrocardiogram (EKG), if indicated
  * Radiologic imaging to evaluate the status of disease may be performed as a part of routine care.
  * Leukapheresis
  * Dendritic cell vaccine preparation
* Procedures during priming vaccination (Days 1 to 3)

  * Complete physical examination (with PS and weight)
  * 19F/1H MRI scanning on day of vaccination, 6 hrs (±1 hour) and 24 hrs (±4 hour) post-injection.
  * Blood for in vitro assays, before first i.d. administration on day 1 (baseline) and after the last i.d. administration on day 3
  * DTH tests: administration on day 1 and readout on day 3
  * Biopsy of the DTH site can be performed in any subject who consented to such biopsy, at the discretion of the investigator/sub-investigator (Day 3 only, based on readout)
* Procedures on Day 15

  * Complete physical examination (with ECOG PS and weight)
  * CBC, platelet, differential
  * Blood for in vitro assays
* Procedures during booster courses (Days 36 to 38, 64 to 66, and 91 to 93)

  * Complete physical examination (with PS and weight) on the 1st day of each 3 day course (Days 36, 64, and 91)
  * CBC, platelet, differential on the 1st day of each 3 day course (Days 36, 64, and 91)
  * Comprehensive metabolic panel (CMP) including: glucose, BUN, creatinine, sodium, potassium, Cl, CO2, calcium, total protein, albumin, alkaline phosphatase, AST, ALT, total bilirubin on the 1st day of each 3 day course (Days 36, 64, and 91)
  * DTH tests: administration on 1st day and readout on 3rd day during 2nd and 3rd booster courses (Administration days 64 and 91, readout days 66 and 93)
  * Biopsy of the DTH site can be performed in any subject who consented to such biopsy, at the discretion of the investigator/sub-investigator (3rd day of 3 day course, based on readout of DTH test)
  * Blood for in vitro assays (1st and 3rd day of each 3 day course)
* Procedures on Day 105

  * Complete physical examination (with ECOG PS and weight)
  * CEA levels in the blood (as a tumor marker)
  * CBC, platelet, differential
  * Comprehensive metabolic panel (CMP) including: glucose, BUN, creatinine, sodium, potassium, Cl, CO2, calcium, total protein, albumin, alkaline phosphatase, AST, ALT, total bilirubin
  * Radiologic imaging to evaluate the status of disease may be performed as a part of routine care
  * Photography
* Long term follow-up The subjects with lack of disease progression at 6 months after the last vaccination will be monitored for the disease free survival and overall survival. Subjects may be contacted every 3 months within the first three years after study intervention, every six months until year 5, and annually afterwards. In lieu of direct contact a medical record review may be performed to obtain the data for these time points for disease progression and/or survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have adequate tumor tissue from surgery, performed as part of their conventional care.
* No chemotherapy, radiotherapy, major surgery, or biologic therapy for their malignancy in the 2 weeks prior to vaccine administration and they must have recovered from all side effects.
* An ECOG performance status of 0, 1, or 2.
* Age equal to 18 years or older.
* Blood tests:

  * Platelet counts greater than 80,000 (platelet count, hematocrit, and WBC will be re-evaluated within 2 weeks prior to leukapheresis)
  * Hematocrit > 27.0
  * White blood count > 2000/µL
  * Creatinine less than or equal to 2 X ULN
* Aware of the neoplastic nature of his/her illness, the experimental nature of the study intervention, alternative treatments, potential benefits and risks, and willing to sign a written informed consent document.

Exclusion Criteria:

* Subjects currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 2 weeks after removal from immunosuppressive treatment. Subjects on maintenance steroids because of adrenal insufficiency are eligible.
* Subjects with total bilirubin greater than 2 X ULN.
* Subjects with uncontrolled pain.
* Subjects with active autoimmune disease, positive serology for HIV, HBV, or HCV. (Hypothyroidism is allowed.)
* Subjects who are allergic to or develop an allergy to heparin.
* Subjects who are pregnant.
* Subjects who have sensitivity to drugs that provide local anesthesia.
* Subjects who have medical contraindications for MRI. Such contraindications include:

  * Electrical implants such as cardiac pacemakers or perfusion pumps
  * Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye or steel implants
  * Ferromagnetic objects such as jewelry or metal clips in clothing
  * Pre-existing medical conditions, including claustrophobic reactions, the likelihood of developing a seizure or any greater than normal potential for cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Adverse events from the labeled DC vaccine | 1 year
Ability to track the labeled DC vaccine by MRI | 1 year

SECONDARY OUTCOMES:
Comparative analysis of the effectiveness of lymph node accumulation of DC vaccines injected to resting versus pre-activated nodes (DCs injected on day 1 versus day 3 of the three day-long vaccination cycle. | 1 year
  Effectiveness of DC accumulation may be correlated with their effectiveness in inducing immune responses as measured by:
  * Increase in the magnitude in the DTH response to: A) autologous tumor lysates (primary endpoint of efficacy); B) KLH; and c) saline (control); all injected intradermally.
  * Peripheral blood CD8+ and CD4+ T cell responses against autologous tumor cells, using IFNγ-ELISPOT readout.
  * In any HLA-A2+ subjects on the protocol, we may evaluate peripheral blood CD8+ T cell responses against CRC-related peptide epitopes present, using IFN ELISPOT as readout.
May assess the disease-free survival and overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David L. Bartlett, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States